CLINICAL TRIAL: NCT03938649
Title: Randomized Phase II Study of Combination Androgen Deprivation Therapy (ADT) and Radiotherapy in High Risk Prostate Cancer: Stereotactic Body Radiotherapy Vs ConventionAl IMRT to Prostate and Pelvic Nodes (SRAM Study)
Brief Title: SRAM Study_Postate Cancer
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: CCTU (Other)
Responsible Party: Sponsor-Investigator, CCTU, Comprehensive Clinical Trial Unit, Chinese University of Hong Kong
Organization: Chinese University of Hong Kong (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: PST008
Record Dates: First submitted 2019-04-18; First posted 2019-05-06 (Actual); Last update posted 2024-12-12 (Actual); Status verified 2024-12

CONDITIONS: Advanced Prostate Cancer

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Conventional IMRT (Experimental): * RapidArc IMRT to prostate and pelvic nodes. 76Gy to prostate, 70Gy to proximal 2/3 of seminal vesicles, and 50Gy to pelvic nodes (up to bifurcation of common iliac nodes).
  * 38 fractions of daily treatment, Monday to Friday
  Interventions: Radiation: Conventional IMRT
- SBRT (Experimental): * RapidArc IMRT to prostate and pelvic nodes. 40Gy to prostate, 36.25Gy to proximal 2/3 of seminal vesicles, and 25Gy to pelvic nodes (up to bifurcation of common iliac nodes)
  * 5 fractions of weekly treatment. Once fraction per week.
  Interventions: Drug: SBRT

INTERVENTIONS:
Radiation: Conventional IMRT — RapidArc IMRT to prostate and pelvic nodes. 76Gy to prostate, 70Gy to proximal 2/3 of seminal vesicles, and 50Gy to pelvic nodes (up to bifurcation of common iliac nodes).
  38 fractions of daily treatment, Monday to Friday.
  All patients will be given neoadjuvant and adjuvant androgen deprivation therapy.
  Arms: Conventional IMRT
Drug: SBRT — RapidArc IMRT to prostate and pelvic nodes. 40Gy to prostate, 36.25Gy to proximal 2/3 of seminal vesicles, and 25Gy to pelvic nodes (up to bifurcation of common iliac nodes) 5 fractions of weekly treatment. Once fraction per week. All patients will be given neoadjuvant and adjuvant androgen deprivation therapy.
  Arms: SBRT

SUMMARY:
This is a phase 2 randomized study for High risk localized prostate cancer (T3 to T4 disease and/or PSA > 20 and/or Gleason score ≥ 8) without evidence of distant and nodal metastasis.

Patient will be randomized to:Arm 1

* Conventional IMRT RapidArc IMRT to prostate and pelvic nodes. 76Gy to prostate, 70Gy to proximal 2/3 of seminal vesicles, and 50Gy to pelvic nodes (up to bifurcation of common iliac nodes).
* 38 fractions of daily treatment, Monday to Friday

or Arm 2

SBRT

* RapidArc IMRT to prostate and pelvic nodes. 40Gy to prostate, 36.25Gy to proximal 2/3 of seminal vesicles, and 25Gy to pelvic nodes (up to bifurcation of common iliac nodes)
* 5 fractions of weekly treatment. Once fraction per week. All patients will be given neoadjuvant and adjuvant androgen deprivation therapy (detail as below)

ELIGIBILITY:
Inclusion Criteria:

* Histological confirmation of prostate adenocarcinoma
* High risk prostate cancer patients (i.e. T3 to T4 disease and/or PSA > 20 and/or Gleason score ≥ 8)
* ECOG performance score 0-1
* Age ≥ 18
* History/physical examination within 2 weeks prior to registration
* Able to sign informed-consent

Exclusion Criteria:

* Patients with active cancer other than prostate cancer and non-melanoma skin cancer.
* Evidence of distant metastases
* Regional lymph node involvement
* Previous radical surgery (prostatectomy), cryosurgery, or HIFU for prostate cancer
* Previous pelvic irradiation, prostate brachytherapy, or bilateral orchiectomy
* Previous hormonal therapy, such as LHRH agonists (e.g., goserelin, leuprolide) or LHRH antagonists (e.g., degarelix), anti-androgens (e.g., flutamide, bicalutamide), estrogens (e.g. DES), or surgical castration (orchiectomy)
* Unstable angina and/or congestive heart failure requiring hospitalization, transmural myocardial infarction within the last 6 months, acute bacterial or fungal infection requiring intravenous antibiotics, chronic obstructive pulmonary disease exacerbation or other respiratory illness requiring hospitalization or precluding study therapy at the time of registration
* Patients who have received prior chemotherapy.

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes
Enrollment: 120 (Estimated)
Dates: Start 2019-05-15 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
To compare acute toxicities between SBRT and conventional IMRT | 4 years
  Toxicities will be assessed by AE CTC version 4 between 2 treatment arms

SECONDARY OUTCOMES:
To compare health-related quality of life (HRQOL) between SBRT and conventional IMRT | 4 years
  Questionnaire EPIC will be used at pre-treatment, during treatment and at 3, 6, 9, 12, 18 and 24 months post treatment
To compare the biochemical-failure free survival at 5 years | 5 years
To compare the progression-free survival at 5 years | 5 years
To compare the overall survival at 5 years | 5 years
To compare the late toxicities between 2 treatment arms | 5 years
  Toxicities will be assessed by AE CTC version 4 between 2 treatment arms

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Clinical Oncology, Prince of Wales Hospital, Hong Kong, Hong Kong

IPD SHARING:
Plan to Share IPD: No